CLINICAL TRIAL: NCT02098759
Title: Long-term, Prospective Study Evaluating Clinical and Molecular Biomarkers of Epileptogenesis in a Genetic Model of Epilepsy - Tuberous Sclerosis Complex
Acronym: EPISTOP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sergiusz Jozwiak (Other)
Collaborators: University of Rome Tor Vergata (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Vrije Universiteit Brussel (Other); General University Hospital, Prague (Other); Charite University, Berlin, Germany (Other); KU Leuven (Other); Medical University of Vienna (Other); Rudolf Magnus Institute - University of Utrecht (Other); Brigham and Women's Hospital (Other)
Responsible Party: Sponsor-Investigator, Sergiusz Jozwiak, MD, PhD, Children's Memorial Health Institute, Poland
Organization: Children's Memorial Health Institute, Poland (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: EPISTOP; 602391 (Other Grant/Funding Number: European Commission, 7th Framework Programme)
Record Dates: First submitted 2014-03-25; First posted 2014-03-28 (Estimated); Last update posted 2014-04-04 (Estimated); Status verified 2014-04

CONDITIONS: TSC; Tuberous Sclerosis Complex; Epilepsy
Keywords: TSC; tuberous sclerosis complex; epilepsy
MeSH Terms: conditions — Tuberous Sclerosis; Epilepsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- epilepsy early diagnosis (Experimental): Infants that have epileptiform discharges on vEEG and no clinical seizures, if their parents/caregivers give consent, will enter the randomized part of the study. Those children will be randomized into two groups: group A will be diagnosed as having epilepsy after subclinical (electroencephalographic) epileptiform discharges, and the patients in group B will be diagnosed as epileptic after clinical seizures appear. All infants diagnosed with epilepsy will receive standard therapy with recommended first line antiepileptic drug starting from the day of diagnosis.
  Interventions: Device: epilepsy early diagnosis protocol
- standard epilepsy diagnosis (Experimental): Infants that have epileptiform discharges on vEEG and no clinical seizures, if their parents/caregivers give consent, will enter the randomized part of the study. Those children will be randomized into two groups: group A will be diagnosed as having epilepsy after subclinical (electroencephalographic) epileptiform discharges, and the patients in group B will be diagnosed as epileptic after clinical seizures appear. All infants diagnosed with epilepsy will receive standard therapy with recommended first line antiepileptic drug starting from the day of diagnosis.
  Interventions: Device: epilepsy early diagnosis protocol

INTERVENTIONS:
Device: epilepsy early diagnosis protocol — Infants that have epileptiform discharges on vEEG and no clinical seizures, if their parents/caregivers give consent, will enter the randomized part of the study. Those children will be randomized into two groups: group A will be diagnosed as having epilepsy after subclinical (electroencephalographic) epileptiform discharges (based on epilepsy early diagnosis protocol), and the patients in group B will be diagnosed as epileptic after clinical seizures appear. All infants diagnosed with epilepsy will receive standard therapy with recommended first line antiepileptic drug starting from the day of diagnosis.

SUMMARY:
The primary objective of clinical part of EPISTOP project is to identify the clinical and molecular biomarkers of epileptogenesis in a prospective clinical study of patients with TSC.

Secondary objective of the clinical part of EPISTOP is to compare the effects of standard antiepileptic treatment in patients diagnosed as having epilepsy after clinical seizures vs after electroencephalographic epileptiform discharges, in a randomized trial in TSC patients.

DETAILED DESCRIPTION:
Overview of study design This is a prospective study of epileptogenesis in TSC infants. In control subjects only one blood sampling will be performed and those infants will not be observed prospectively.

The study consists of two phases: (1) prospective tracking of epileptogenesis by means of serial vEEG recordings; (2) treatment of epilepsy diagnosed after clinical or after electroencephalographic epileptiform discharges.

All patients enrolled in the study will participate in the first phase. The second phase will concern only the children with epilepsy with electroencephalographic epileptiform discharges and/or clinical seizures, whose parents/caregivers will give consent for the randomized part of the project.

At baseline, all patients will undergo neuroimaging examination by means of MRI, a battery of neuropsychological tests, blood biomarker sampling, and the review of medical history of the patient and the family.

Epileptogenesis in TSC infants will be tracked by means of serial vEEG recordings. In children with diagnosed epilepsy, standard therapy with recommended first line antiepileptic drug will be given. Children with clinical seizures, either noticed by a caregiver, or a treating neurologist or recorded on video during vEEG will be immediately diagnosed as having epilepsy. Infants that have epileptiform discharges on vEEG and no clinical seizures, if their parents/caregivers give consent, will enter the randomized part of the study. Those children will be randomized into two groups: group A will be diagnosed as having epilepsy after subclinical (electroencephalographic) epileptiform discharges, and the patients in group B will be diagnosed as epileptic after clinical seizures appear. All infants diagnosed with epilepsy will receive standard therapy with recommended first line antiepileptic drug starting from the day of diagnosis.

Children whose parents/caregivers will not give consent for the randomized part of the project, will be followed with serial vEEG and epilepsy will be diagnosed after clinical seizures.

Children without seizures and no epileptiform discharges on vEEG will be followed without treatment.

Blood samples for biomarker studies will be collected at study entry, at the onset of epileptiform discharges on vEEG or at the age of 6 months, whichever is applicable, at the onset of clinical seizures, and at the end of follow-up (age 2 years) in all patients participating in the project.

At the age of 24 months, all TSC infants participating in the study will undergo neuroimaging examination by means of MRI, a battery of neuropsychological tests, and epilepsy analysis.

Statistical considerations Full analysis set comprises all patients participating in the study, including the control group. This set will be divided into subsets: control group, TSC patients with epilepsy, and TSC patients with no epilepsy. Among TSC patients with epilepsy, patients with well-controlled seizures and patients with drug-resistant epilepsy will be identified. In full analysis set the blood biomarkers will be analysed. Clinical analysis set will comprise of all TSC infants enrolled in the study and the clinical biomarkers of epileptogenesis (neuroimaging, vEEG, data from medical history) will be analysed in this set. Treatment analysis set will comprise of infants participating in the randomized part of the study and the efficacy of antiepileptic treatment in respect to the point of epilepsy diagnosis (electroencephalographic epileptiform discharges onset in group A and clinical seizures onset in group B) will be assessed in this set.

The interim analyses will be performed when 70% of the patients will complete the whole study. Final analyses will be performed when the last patient will complete the study (at the age of 24 months).

Rationale for the study design This study is composed of two phases: (1) prospective tracking of epileptogenesis by means of serial vEEG recordings; (2) treatment of epilepsy diagnosed after clinical or after electroencephalographic epileptiform discharges. All TSC infants enrolled in the study as well as control children will participate in phase 1, whereas only children diagnosed with epilepsy will participate in phase 2. The time point of epilepsy diagnosis (at the onset of electroencephalographic epileptiform discharges or clinical seizures) will be randomly assigned to participating children by central randomizer and will be blinded to the patients' caregivers and treating neurologists.

The identification of the biomarkers of ongoing epileptogenesis, as well as delineation of the point of no return, at which the occurrence of clinical seizures is inevitable, requires the prospective study, starting before the onset of clinical seizures. To achieve the clinical usefulness of potential biomarkers, they should be based on the analysis of standard clinical tests: neuroimaging by means of MRI, EEG, blood samples.

Our study will use the standard clinical tests to identify the biomarkers of epileptogenesis on neuroimaging studies, EEG, and in the blood samples in TSC infants before and after the onset of seizures, to track the changes in measured parameters during ongoing epileptogenesis. Investigators will compare the results obtained in individual patients before the onset of EEG abnormalities, after the onset of electroencephalographic epileptiform discharges, after clinical seizures and at the age of 24 months. In order to identify the risk of epilepsy among TSC patients, Investigators will compare the results obtained in patients who develop epilepsy and those who remain epilepsy free. We will also compare the results obtained in TSC children with age-matched non-epileptic infants.

The aim of the study is to establish the earliest possible point to diagnose epilepsy in TSC infants. It is now widely accepted that the clinical seizures are preceded by the progressing deterioration of EEG. Such deterioration is not seen in TSC infants who do not develop clinical seizures. EEG is a standard, non-invasive procedure in epileptic children. Therefore, EEG will be used to track epileptogenesis and to set the points for biomarkers sampling. Patients with epileptiform discharges on EEG recordings will enter the blinded, randomized part of the study, aimed to compare the effects of preclinical diagnosis and treatment of epilepsy vs diagnosis and treatment after clinical seizures appearance.

To ascertain blinding of the study, the reports of vEEG recordings will not be sent to treating neurologist, but only to central randomizer. He will provide the treating neurologist with the diagnosis of epilepsy or no epilepsy, without giving the details of EEG. If the diagnosis of epilepsy is provided, it can mean either of the following: the patient had clinical seizures recorded on videoEEG, or had electroencephalographic epileptiform discharges and was randomized to group diagnosed with epilepsy at that point. Similarly, if the treating neurologist receives a diagnosis of no epilepsy in a patient, it is not known whether EEG was normal, or the patient had epileptiform EEG, but was randomized to group diagnosed as epileptic at the onset of clinical seizures.

Taken together, the treating neurologist and the patient's parents/caregivers will be blinded to the diagnostic approach in a patient, but at the same time, an adequate treatment can be implemented.

Epileptiform discharges on EEG not only precede clinical seizures, but also reflect changes in the brain that may per se cause neurodevelopmental delay and autism in children. In animal models it was shown that epileptogenesis could be interfered by antiepileptic treatment implemented before the onset of clinical seizures. A recent study showed that initiation of antiepileptic treatment before the onset of clinical seizures but after the onset of epileptiform discharges on EEG reduced the risk of mental retardation and drug-resistant epilepsy. Amelioration of epilepsy by implementation of antiepileptic drugs before the clinical seizures onset was also shown in neonates with severe hypoxic-ischemic encephalopathy. Current guidelines for epilepsy management in TSC patients recommend treatment of subclinical seizures equally to standard treatment after clinical seizures onset.

Patients' numbering Each patient will be identified in the study by code, that will be assigned during baseline visit. This code will be the primary identifier of the patient throughout the study. The code will consist of site identifier and sequential patient number (for example: 01-001). Once assigned, the patient's code cannot be re-used or changed.

Randomization procedures Patients with epileptiform discharges on vEEG noted prior to clinical seizures will enter the randomized part of the study. The time point of randomization will not be known to the treating neurologist to keep the study blinded. Central randomizer will provide the diagnosis of the patient to the treating neurologist after each EEG recording.

Randomization will be performed as block randomization stratified for centre. Patients will be randomized in ratio 1:1.

Adverse events An Adverse Event (AE) is any adverse change from the patient's baseline condition that occurs during the course of the study, irrespective to the relation to the epilepsy approach. However, it is important that this study does not test any investigational product, so only the undesirable effects of epilepsy diagnosis before or after the onset of clinical seizures should be considered as study-related (and not drug-related, as there is no investigational drug).

Adverse events do not include:

* epileptic seizures, unless worsened due to late epilepsy diagnosis;
* planned medical or surgical procedures, ie. vaccinations, hospitalizations related to control examinations, like cardiologic follow-ups etc.
* pre-existing disease or medical condition that does not worsen, However, these events should be mentioned in eCRF (in Others or Comments section in the respective visit record). Seizures must be reported on dedicated eCRF sections. Parents of patients experiencing seizures should be asked to report the number and type of seizures daily and these data should be transferred to eCRF.

For each AE, the relation to the study should be assessed by the investigator and reported in eCRF. If the causal relationship between the AE and the project is possible or certain, the relevant comment including the justification must be recorded on eCRF.

Serious Adverse Events (SAE) is any AE fulfilling any of the following criteria:

* fatal
* life-threatening
* requiring hospitalization or prolongation of existing hospitalization, with the exception of planned hospitalizations
* resulting in persistent or significant disability
* medically significant or requiring intervention to prevent any of the outcomes listed above All SAE regardless their relation to the study must be recorded in eCRF and reported to the Project Coordinator (Sergiusz Jóźwiak, at IPCZD) within 48 hours by fax: +48 22 815 74 02 or e-mail: sergiusz.jozwiak@gmail.com The coordinator will contact appropriate health authorities as well as Scientific Advisory Board and Ethics Committee. All SAEs must be followed until resolution or stabilization. Follow up report must be recorded within 30 days after the onset of SAE or earlier, if possible, and reported to the Study Coordinator by fax or e-mail.

Data collection and management Clinical data will be captured using electronic Case Report Form (eCRF). Data will be documented in various source documents and then manually entered into the eCRF by study site personnel. eCRF will be provided to each site by IPCZD.

All information about study subjects will be confidential and managed according to local regulations and laws. Specifically, a signed authorization of the patient's caregivers informing of the following is required:

* what protected health information will be collected from the patients in this study
* who will have access to that information and why
* who will use or disclose that information
* the rights of the study subject caregivers to revoke their authorization for use of their protected health information.

The patient's caregivers will be told that representatives of the Consortium, ethics committees, and regulatory authorities may inspect their medical records to verify the information collected. They will also be told that all personal data available for the inspection will be handled in strictest confidence and in accordance with local data protection laws.

In case that a patient's caregivers revoke their authorization to use or to collect protected health information, only information collected prior to the revocation of the authorization can be used.

Following the study completion, all documents related to the project, including patients' source data, should be stored on site according to local legal regulations.

Monitoring plan Monitoring will be performed by monitor (CRA) chosen by IPCZD, coordinating site. In each participating centre one monitoring visit will be conducted annually.

Verification of source data

* 100% check of presence and correctness of Informed Consent Forms
* 100% check of inclusion and exclusion criteria
* 50% check of source documents of the following study data:

  * Age
  * Sex
  * Diagnosis TSC
  * Diagnosis allocation
  * Date of inclusion
  * Result of MRI, EEG and neuropsychological tests
  * Seizures diary
* 100% check of SAE's and SUSAR's as well as verification of the appropriate reporting procedures General control
* For each visit of each centre the rate of inclusion and the dropout rate will be reported.
* For each centre the presence and completeness of the Investigator Site File will be checked and for the sponsor the Trial Master File will be checked as well.
* For each centre study procedures will be checked as well as the ability of the study personnel to comply with these procedures.

Reporting The monitor will provide a written report to the sponsor after each visit to a study location. This report will be stored by the sponsor and will be directly available for an audit. A study location will receive a written summary of the control procedures that have been performed and the associated findings.

The 'monitor visit report' will include:

* A summary of control procedures performed by the monitor
* A general description of quality at the study site
* A summary stating the most important findings / facts, deviations and shortcomings
* An overview of proposed measures and recommendations to ensure compliance with the protocol
* The general conclusion The sponsor will receive the originals of initiation visit report and the close-out visit report and principal investigator of each site will receive copies of these documents. If applicable, other relevant contacts considering the trial will be enclosed as a written report.

Data quality assurance The eCRFs and other essential documents will be reviewed by a clinical monitor designed by IPCZD.

Essential documents include:

* signed informed consent documents for all subjects
* the decision of ethics committee together with the composition of ethics committee
* records of all communications between the investigator and the ethics committee
* all source documents (patient records, hospital records, laboratory records, seizure diaries, etc)
* any other documents required by local laws or GCP guidelines. Data on CRFs will be source-verified during site visits for accuracy and completeness according to the monitoring plan. The visits will take place annually as the minimum. The first visit will be scheduled 12 months after the first visit of the first patient enrolled by the site. The investigator will allocate adequate time for such monitoring activities. The investigator will also ensure that the monitor is given access to all above noted study documents and has adequate space to conduct the monitoring visit.

The safety of patients in the study will be monitored by Independent Ethics Board supported by a biostatistician designated by IPCZD. The Independent Ethics Board will perform the review of the safety and efficacy after 70% of all planned randomized patients complete the study and their seizures outcome data are available.

Early stopping rules The randomized part of the study can be stopped early if the external Scientific Advisory Board together with Steering Committee decides so, based on the analysis of study safety and/or efficacy. Particularly, the study can be stopped for unacceptable safety. In this case, all participating and new patients will enter the observational part of the project only.

Second, the study may be stopped if any of the compared epilepsy approaches (early diagnosis versus diagnosis after clinical seizures) shows clear benefit in terms of seizure outcome, evidenced by the interim statistical analysis. Seizure outcome includes the number of seizure-free patients, the number of patients with normalized EEG, and the number of patients with drug-resistant epilepsy. The interim analysis will be performed when 70% of all planned randomized patients complete the study and their seizures outcome data are available. The statistical significance of P-value of 0.001 at interim analysis as evidence to stop early for benefit is required. In this case, all new patients and patients already participating in the study but not having abnormal EEG yet, will be offered the approach that was proved to be significantly more efficient. Other patients already participating in the study will continue their treatment.

Withdrawal of individual subjects Subjects can leave the study at any time for any reason if they wish to do so without any consequences. The investigator/ treating physician can decide to withdraw a subject from the study whenever he/she considers that continuation in the trial would adversely affect the subjects' health. Participants that are under follow-up and treatment of the collaborating centres will continue to be so.

Statistical analyses Full analysis set comprises all patients participating in the study, including the control group. This set will be divided into subsets: control group, TSC patients with epilepsy, and TSC patients with no epilepsy. Among TSC patients with epilepsy, patients with well-controlled seizures and patients with drug-resistant epilepsy will be identified. In full analysis set the blood biomarkers will be analysed. Clinical analysis set will comprise of all TSC infants enrolled in the study and the clinical biomarkers of epileptogenesis (neuroimaging, vEEG, data from medical history) will be analysed in this set. Treatment analysis set will comprise of infants participating in the randomized part of the study and the efficacy of antiepileptic treatment in respect to the point of epilepsy diagnosis (electroencephalographic epileptiform discharges onset in group A and clinical seizures onset in group B) will be assessed in this set.

The interim analyses will be performed when 70% of the patients will complete the whole study. Final analyses will be performed when the last patient will complete the study (at the age of 24 months).

Regarding clinical outcome measures and the study endpoints, the sample size was determined based on our previous study, in which similar parameters were assessed. The statistical analysis will include two types of tests:

* qualitative variables (frequencies of occurrence) will be analysed using chi-square tests
* quantitative variables using non-parametric equivalencies of ANOVA tests. The power of these tests was calculated for the p-level (alpha error) set at 0.5, and assuming the balanced distribution of patients in the groups. As described, we expect that 60-70% of subjects will have subclinical seizures prior to onset of clinical epilepsy, and thus be randomized to either A or B group. We predict that early diagnosis and treatment will be 50-60% effective in preventing clinical seizure development in the patients that are randomized to group A. Given a set of 60 patients, with 30 going to group A and 30 to group B, our power to detect this difference in clinical seizure development is higher than 80%. All calculations were done using G*Power v 3.1.3 freeware, Kiel University, Germany.

Ethical considerations

EPISTOP project was designed and shall be implemented and reported in accordance with ICH Harmonized Tripartite Guidelines for Good Clinical Practice and the following EU legislations:

* The Charter of Fundamental Rights 2000 of the EU;
* European Directives 95/46/EC, 2002/58/EC, and 2001/20/EC.

All participants in EPISTOP will respect the ethical principles laid down by national regulations and the following international conventions and declarations:

* Helsinki Declaration;
* Oviedo Convention of the CE on Human Rights and Biomedicine;
* UN Convention on the Rights of Child;
* Universal Declaration on the human genome and human rights adopted by UNESCO. This clinical study was designed, shall be implemented and reported in accordance with Good Clinical Practice, the regulations given in EU Directive No 20/2001 and other relevant regulations to ensure patients' safety. All Investigators will use a unified electronic Case Report Form to ensure the quality of data entered into the database, and an external data monitor (Clinical Research Associate; CRA) to monitor the progress of the study. Ethics issues will be supervised also by the external Scientific Advisory Board and Ethical Committee.

EPISTOP has been already accepted by the local Ethics Boards at the Children's Memorial Health Institute (IPCZD), at Universita Degli Studi Di Roma Tor Vergata (TVG) and at Fakultni Nemocnice V Motole (UHM).

Personal data protection EPISTOP will follow the principles for the protection of personal data laid down by European legal regulations. The study coordinator will ensure that consent for data storage is obtained from all participants and the data will be used only if there is consent for its use. Study subjects genetic, epigenetic, biochemical, proteomic, electroencephalographic, neuroimaging, and other medical data will be stored and analyzed in a coded/anonymous form. Data management and data safety reports will be regularly presented to the Advisory Board.

Electronic case report form will be used for web-based data entry. The data entered into this database will be de-identified and only the responsible researchers will have the access to identifying details.

The collaborative nature of EPISTOP requires the exchange of information and biological material between European and US partners. For purposes of WP3, WP5, WP7, biological samples obtained from patients and the relevant medical data will be transferred between sites. Only de-identified and coded samples as well as necessary medical data will be sent. The special safety provisions concerning biological material transportation will be considered and has been taken into account when calculating the costs of the project.

The participants of EPISTOP and/or their legal representatives will be informed that they have the right to cancel their consent at any time by giving written notice to investigator. If the consent is cancelled, then the investigators will no longer use or disclose any medical information of the participant. However, canceling this consent will not affect previous uses and disclosures and the already existing participant's medical information would not be removed from the study records.

The data produced in this study will be stored in a locked, secure location. Only members of the research team will have access to this location. Following completion of the research study the data will be kept as long as required by law and then destroyed as required by the hospital, laboratory or institute policy.

EPISTOP assures that the key design elements of the project will be posted in its publicly accessible website. The results of the project will be submitted to publication in medical journals with the respect of participants' personal data protection.

ELIGIBILITY:
Inclusion criteria

Inclusion criteria for TSC patients:

* male or female infants with a definite diagnosis of TSC (Roach criteria; Roach 1998 or DNA confirmed),
* age up to 4 months at the moment of enrolment,
* no clinical seizures seen by caregivers or on baseline videoEEG recording,
* written informed consent of caregivers. It is possible to give consent for the observational part of the study only. In this case, the child will not enter the randomized part of the study.

Inclusion criteria for the control group:

* male or female infants who have undergone routine MRI for reasons other than epilepsy and brain tumor or cortical defects,
* age up to 24 months at the moment of study entry,
* written informed consent of caregivers. Exclusion criteria

Exclusion criteria for TSC patients:

* any type of seizures observed till baseline visit,
* antiepileptic treatment at or prior to study entry,
* contraindications to MRI,
* any severe and/or uncontrolled medical condition that is considered by the investigator as possibly affecting the EPISTOP analyses or procedures.

Exclusion criteria for the control group:

* any sign or symptom suggesting TSC diagnosis,
* any type of seizures observed at study entry,
* antiepileptic treatment at study entry,
* history of seizures, with the exception of febrile seizures,
* any severe and/or uncontrolled medical condition that is considered by the investigator as possibly affecting the EPISTOP analyses or procedures.

Max Age: 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2013-11; Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
number of patients with epilepsy | at 24 month of life
  Full analysis set comprises all patients participating in the study, including the control group. This set will be divided into subsets: control group, TSC patients with epilepsy, and TSC patients with no epilepsy. Among TSC patients with epilepsy, patients with well-controlled seizures and patients with drug-resistant epilepsy will be identified. In full analysis set the blood biomarkers will be analysed. Clinical analysis set will comprise of all TSC infants enrolled in the study and the clinical biomarkers of epileptogenesis (neuroimaging, vEEG, data from medical history) will be analysed in this set. Treatment analysis set will comprise of infants participating in the randomized part of the study and the efficacy of antiepileptic treatment in respect to the point of epilepsy diagnosis (electroencephalographic epileptiform discharges onset in group A and clinical seizures onset in group B) will be assessed in this set.

CONTACTS AND LOCATIONS:
Overall Officials: Seriusz Jozwiak, Md, PhD, Principal Investigator — Children's Memorial Health Institute
Locations (9):
- Medizinische Universitaet Wien, Vienna, Austria
- Belgium (2):
  - Vrije Universiteit Brussel, Brussels
  - Katholieke Universiteit Leuven, Leuven
- Fakultni Nemocnice V Motole, Prague, Czechia
- Institut National De La Sante et de la Recherche Medicale, Paris, France
- Charite - Universitaetsmedizin Berlin, Berlin, Germany
- Universita Degli Studi Di Roma Tor Vergata, Rome, Italy
- Universitair Medisch Centrum Utrecht, Utrecht, Netherlands
- Children's Memorial Health Institute, Warsaw, Poland

REFERENCES:
- [Derived] van der Poest Clement E, Jansen FE, Braun KPJ, Peters JM. Update on Drug Management of Refractory Epilepsy in Tuberous Sclerosis Complex. Paediatr Drugs. 2020 Feb;22(1):73-84. doi: 10.1007/s40272-019-00376-0. PMID 31912454